CLINICAL TRIAL: NCT07191522
Title: Efficacy of Photodynamic Therapy in the Non-Surgical Treatment of Peri-Implantitis
Acronym: PeriimpMAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aPDT MAA; Research Grant (Other: Egas Moniz School of Health and Science)
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Peri Implantitis
Keywords: Peri-implantitis; Antimicrobial Photodynamic Therapy
MeSH Terms: conditions — Peri-Implantitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Mechanical debridment with titanium curettes and ultrasounds
  Interventions: Procedure: Mechanical debridment with titanium curettes and ultrasounds
- Study Group (Experimental): Mechanical debridment with titanium curettes and ultrasounds + aPDT (antimicrobial photodynamic therapy)
  Interventions: Procedure: Mechanical debridment with titanium curettes and ultrasounds + aPDT (antimicrobial photodynamic therapy)

INTERVENTIONS:
Procedure: Mechanical debridment with titanium curettes and ultrasounds — Removal of deposits above and below the gum line using hand or ultrasonic tools to reduce the inflammatory parameters
  Arms: Control Group
Procedure: Mechanical debridment with titanium curettes and ultrasounds + aPDT (antimicrobial photodynamic therapy) — Non-invasive treatment that uses a combination of a light-sensitive compound (photosensitizer), specific light and oxygen to generate reactive oxygen species (ROS) that kill bacteria
  Arms: Study Group

SUMMARY:
Peri-implantitis is a growing public health problem that can lead to several complications and sequelae, with a serious impact on the health and quality of life of patients and a high cost for healthcare systems.

Bacterial plaque that accumulates around dental implants leads to peri-implant tissue inflammation that ultimately can result in the loss of the implant, significant bone destruction and infection that can reach other regions. Successful implant decontamination is necessary to preserve the implant and several strategies have been suggested for this purpose, however, there is still no fully effective treatment modality and failures and recurrence are relatively frequent.

To better understand this problem and develop more effective treatment strategies, investigators will first conduct an epidemiological study to understand the factors associated with the development of this pathology. Although there is data at an international level, the incidence of this problem in Portugal has not yet been properly studied. Later investigators will conduct a randomized clinical trial to evaluate the 6-week clinical outcomes of patients treated with a photodynamic therapy as an adjuvant versus the use of conventional titanium implant curettes for implant surface decontamination in the non-surgical treatment. Sixty patients/implants with peri-implantitis and within the established criteria, will undergo non-surgical treatment with one of the two protocols being studied. Various clinical and radiographic parameters will be evaluated, such as probing depth, insertion loss, recession, bleeding on probing, suppuration, peri-implant crevicular fluid volume, alveolar bone loss and peri-implantitis microbiome will be evaluated before surgery and 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age;
* patients with one or more implants diagnosed with peri-implantitis rehabilitated for at least one year;
* PI and GI < 25%.

Exclusion Criteria:

* smoking patients;
* patients with uncontrolled periodontitis;
* systemic diseases that influence the study (diabetes);
* inadequate prosthetic rehabilitation that cannot be modified or that prevents access for physical decontamination;
* implants rehabilitated with cemented crowns;
* pregnant and lactating women;
* previous surgical intervention at the same site;
* therapy with non-steroidal anti-inflammatory drugs (NSAIDs), antibiotics or immunosuppressants in the last 3 months;
* patients previously undergoing chemotherapy or radiotherapy;
* PI and IG > 25%;
* uncooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Probing Depth | From enrollment to the end of treatment at 3 months
  Measuring in milimeters the distance from the gingival margin to the base of a sulcus or peri-implant pocket, using a periodontal probe.

SECONDARY OUTCOMES:
Clinical attachment level | From enrollment to the end of treatment at 3 months.
  Measured with a periodontal probe as the distance from a fixed reference point (usually the implant shoulder or gingival margin) to the base of the peri-implant pocket.
Bleeding on Probing | From enrollment to the end of treatment at 3 months.
  Assessed during gentle probing; bleeding indicates a positive site.
Suppuration | From enrollment to the end of treatment at 3 months.
  Detected by probing or gentle pressure, with purulent exudate confirming presence.
Radiographic bone level | From enrollment to the end of treatment at 3 months.
  Assessed on standardized periapical radiographs, measuring the distance from a fixed reference point (implant shoulder or platform) to the most coronal bone-to-implant contact.
Microbiology outcome | From enrollment to the end of treatment at 3 months.
  Changes in the microbiome collected from peri-implant pockets sequencing 16S ribosomal RNA gene

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Alves, PhD, Principal Investigator — Egas Moniz School of Health and Science
Locations (1):
- Egas Moniz School of Health and Science, Almada, Monte Da Caparica, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LED website — https://www.bredent-implants.com/products-solutions/regeneration/helbo/